CLINICAL TRIAL: NCT03030716
Title: Long-term, Multiple Daily Condensed Tannin Supplementation in Increasing Concentrations Does Not Affect Iron Status or Bioavailability: Results From the Tannin-dose Response Trial.
Brief Title: Multiple Daily Condensed Tannin Supplementation and Iron Bioavailability: The Tannin Dose Response Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Collaborators: United States Department of Agriculture Foreign Agricultural Service (Other)
Responsible Party: Principal Investigator, Brian Lindshield, Ph.D., Associate Professor, Kansas State University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRPTanninTrial
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Iron Deficiency Anemia; Iron-deficiency
Keywords: antinutrients; tannins; proanthocyanidins; salivary proline-rich proteins
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.03 mg 95% condensed proanthocyanidin (Experimental): 0.03 g 95% condensed proanthocyanidins from grape seed extract at week 0 0.03 g 95% condensed proanthocyanidins from grape seed extract at week 4
  Interventions: Dietary Supplement: 95% condensed proanthocyanidins from grape seed extract
- 0.25 g 95% condensed proanthocyanidin (Experimental): 0.25 g 95% condensed proanthocyanidins from grape seed extract at week 0 0.25 g 95% condensed proanthocyanidins from grape seed extract at week 4
  Interventions: Dietary Supplement: 95% condensed proanthocyanidins from grape seed extract
- 1.5 g 95% condensed proanthocyanidin (Experimental): 1.5 g 95% condensed proanthocyanidins from grape seed extract at week 0 1.5 g 95% condensed proanthocyanidins from grape seed extract at week 4
  Interventions: Dietary Supplement: 95% condensed proanthocyanidins from grape seed extract

INTERVENTIONS:
Dietary Supplement: 95% condensed proanthocyanidins from grape seed extract — 0.03, 0.25, and 1.5 g 95% condensed proanthocyanidins from grape seed extract consumed three times daily for 4 weeks each

SUMMARY:
Tannins are known to inhibit iron absorption through formation of insoluble tannin-mineral complexes, and have thus been termed 'antinutritional.' Despite this, there is evidence that adaptation to similar antinutritional factors is possible when consumed over time. Limitations in current studies include short (single meal) duration, and use of incongruent tannin types from the condensed tannins that are commonly consumed. If adaptation to tannins does happen, it may be due to salivary proline-rich proteins, which have been found to be protective of iron status in animal models. The primary objectives of this study are: 1) To determine whether condensed tannins impact iron bioavailability or status when consumed in multi-dose, multiple daily supplements and 2) to test whether salivary protein production may impact iron bioavailability with tannin supplementation. Secondary objectives included assessment of the reliability of astringency as a measure of salivary protein production and iron absorption.

The study has been conducted in an iron absorption study of 11 women, aged 18-35 years old, to determine iron bioavailability with supplementation of 0.03, 0.25, and 1.5 g 95% proanthocyanidin rich grape seed extract before and after regular, three times daily supplementation for four weeks. Each participant consumed all three concentrations of supplement over the 26-week study, with a two-week washout between interventions. Direct iron absorption was measured using area under the curve. Iron status was measured by changes in hemoglobin and ferritin, and was adjusted by participant c-reactive protein levels. Salivary samples were collected before and after supplement consumption during meal challenges, and analyzed on HPLC. Astringency testing was conducted at the end of each meal challenge. Iron absorption and status markers were analyzed by ANOVA, and mixed-modeling followed by pairwise comparison by least significant differences. Pearson's correlations were used to correlated salivary proteins and astringency with iron bioavailability.

The present study will provide important information regarding the approximate influence of condensed tannin consumption on iron bioavailability and storage over time, at different doses. Data will also help to delineate possible physiological mechanisms underlying tannin adaptation and possible ways to detect individuals who better adapt than others.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18-35 years old
* Non-obese BMI (18-29.9)
* Signed informed consent

Exclusion Criteria:

* Oral disease
* Gastrointestinal disease
* Tobacco user
* Heavy alcohol user
* Pregnancy (assessed by pregnancy test)
* Lactation
* Medications affecting iron bioavailability
* Vitamin or mineral supplementation (other than vitamin B12)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2016-06-25 (Actual); Primary Completion 2016-12-10 (Actual); Study Completion 2016-12-10 (Actual)

PRIMARY OUTCOMES:
Change in baseline to endline area under the curve after meal challenge at weeks 0 and 4 of each intervention | Baseline and 4 weeks
  Change in area under the curve will be measured after administration of test meal including ferrous sulfate and condensed tannin supplementation at weeks 0 and 4
Change in baseline to endline hemoglobin and serum ferritin at weeks 0 and 4 of each intervention | Baseline and 4 weeks
  Change in ferritin and hemoglobin will be measured before administration of test meals at weeks 0 and 4
Change in salivary proteins at weeks 0 and 4 of each intervention | Baseline and 4 weeks
  HPLC determination of salivary proteins will be analyzed from saliva collected before and after test meals at weeks 0 and 4 of each intervention

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Lindshield, Ph.D., Principal Investigator — Kansas State University
Locations (1):
- Physical Activity and Nutrition Research Consortium, Manhattan, Kansas, United States

IPD SHARING:
Plan to Share IPD: No